CLINICAL TRIAL: NCT06351800
Title: Universal Prevention of Depression and Anxiety in the General Population Through a Personalized Intervention Based on Risk Algorithms, ICTs, and Decision Support Systems: Randomized Controlled Trial. The "PredictPlusPrevent" Study
Brief Title: The PredictPlusPrevent Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Mediterranean Institute for the Advance of Biotechnology and Health Research (Other)
Responsible Party: Principal Investigator, Juan Ángel Bellón, Principal Investigator, The Mediterranean Institute for the Advance of Biotechnology and Health Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PE-0280-2018
Record Dates: First submitted 2024-03-25; First posted 2024-04-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Depression; Anxiety Disorders
Keywords: Depression; Anxiety Disorders; Prevention; m-health; App; Randomized Controlled Trial
MeSH Terms: conditions — Depression; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Predictplusprevent intervention (Experimental): The intervention will provide information about the likelihood of experiencing depression and anxiety. Additionally, it will offer a personalized depression prevention plan (PPP) based on various interventions such as physical exercise, sleep, expanding relationships, problem-solving, improving communication, assertiveness, decision-making, and managing thoughts.
  Interventions: Behavioral: Predictplusprevent intervention
- Active control group (Active Comparator): The intervention in the active control group will involve assessing the risk level of experiencing depression and/or anxiety in the next 12 months every 3 months. Additionally, participants assigned to this intervention will have free access to the 24 self-help booklets for preventing depression and anxiety included in the 'predictplusprevent' web platform. However, this group will not receive personalized prevention plans, decision support systems, or monitoring and feedback. They will also not have access to the 8 self-guided and interactive modules used in the intervention group.
  Interventions: Other: Psychoeducational intervention

INTERVENTIONS:
Behavioral: Predictplusprevent intervention — The intervention is based on validated risk algorithms to predict depression and anxiety and includes: 1) Mobile applications as main user's interface; 2) a DSS that helps participants to develop their own personalized plans to prevent (PPP) depression and/or anxiety; 3) eight intervention modules (the core of the system) including activities to prevent depression and anxiety, to be proposed and monitoring by the DSS. The intervention is biopsychosocial and multi-component, including the following modules: physical exercise, improving sleep, expanding relationships, problem solving, improving communication skills, assertiveness training, making decisions and managing thoughts. Participants will implement the recommendations and the tool will monitor these actions, offering feedback to improve their PPP at 3, 6, 9 and 12 months.
  Arms: Predictplusprevent intervention
Other: Psychoeducational intervention — To know the level of risk of experiencing depression and/or anxiety in the next 12 months. In addition, participants assigned to this intervention will have free access to the 24 self-help pamphlets for preventing depression and anxiety.
  Arms: Active control group

SUMMARY:
Objective: To design, develop, and evaluate a personalized intervention for the universal prevention of depression and anxiety in the general population based on risk algorithms, ICTs, and decision support systems (DSS).

Methods: A double-blind, parallel-group, randomized controlled trial with a twelve-month follow-up. The entire process of recruitment, random allocation, intervention, and follow-up will be conducted through the 'PredictPlusPrevent' platform and its associated apps. Following a media campaign, at least 9,000 Spanish participants aged 18 to 55 years without depression and/or anxiety at baseline will be randomly assigned to the intervention or active control group "PredictPlusPrevent". The "PredictPlusPrevent" intervention will be self-guided and implemented through participants' smartphones via an app; it will have a biopsychosocial and multi-component approach (8 modules: physical exercise, improving sleep, expanding relationships, problem-solving, improving communication, assertiveness, decision-making, and managing thoughts). The "PredictPlusPrevent" intervention is based on validated risk algorithms for depression and anxiety and a DSS that will help participants develop their own personalized depression prevention plans, which they will implement themselves while the platform monitors and provides feedback. The active control "PredictPlusPrevent" will include information from the risk algorithms and 24 self-help booklets. The primary outcome will be the incidence of new cases of depression and/or anxiety assessed using the PRIME-MD questionnaire, and secondary outcomes will include reductions in depression (PHQ-9) and anxiety symptoms (GAD-7), probability of depression and anxiety risk (predictD and predictA algorithms), and physical and mental quality of life (SF-12).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years.
* Participants must have a smartphone for their own use in the next year.

Exclusion Criteria:

* Not signing the informed consent.
* Having depression and/or anxiety at baseline according to the PRIME-MD questionnaire.
* Living outside of Spain.
* Having a severe mental disorder (psychosis, bipolar disorder, addictions, etc.), a terminal illness or cognitive impairment (dementia).
* Difficulties in understanding Spanish.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9000 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-03-07 (Estimated); Study Completion 2028-03-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of depression and/or anxiety disorders. | 12 months
  Incidence of depression and/or anxiety disorders by Primary Care Evaluation of Mental Disorders (PRIME-MD). PRIME-MD is a diagnostic tool to diagnose depression and anxiety disorders.

SECONDARY OUTCOMES:
Depressive symptoms measured by the Patient Health Questionnaire-9 (PHQ-9). | 12 months
  The Patient Health Questionnaire-9 (PHQ-9) measures symptoms of depression through 9 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of depression, the scalen range is 0 to 27 (9 items).
Anxious symptoms measured by the General Anxiety Questionnaire (GAD-7). | 12 months
  The General Anxiety Questionnaire (GAD-7) measures generalized anxiety disorder through 7 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of anxiety, the scale range is 0 to 21 (7 items).
Probability of depression measured by the Spanish predictD risk algorithm. | 12 months
  The Spanish predictD risk algorithm measures 13 risk factors for depression.
Probability of anxiety measured by the Spanish predictA risk algorithm. | 12 months
  The Spanish predictA risk algorithm measures 12 risk factors for anxiety disorders.
Quality of life measured by the 12-item Short Form (SF-12). | 12 months
  The 12-item Short Form (SF-12) measures quality of life related to physical health and quality of life related to mental health. Scores on the scales range from 0 to 100. Higher scores are equivalent to better health-related quality of life.

IPD SHARING:
Plan to Share IPD: Undecided